CLINICAL TRIAL: NCT00828581
Title: An Open-Label, Single-Dose Study of the Pharmacokinetic Properties of Lorcaserin in Obese or Overweight Elderly Subjects
Brief Title: Pharmacokinetic Properties of Lorcaserin in Obese or Overweight Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APD356-018
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2009-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorcaserin (Experimental)
  Interventions: Drug: lorcaserin

INTERVENTIONS:
Drug: lorcaserin

SUMMARY:
The purpose of this study is to evaluate the PK properties of lorcaserin in obese or overweight elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females
2. Control (Adult) group: aged between 18 and 65 years (inclusive)
3. Elderly group: aged > 65 years (includes subjects 1 day or more beyond the 65th birthday)
4. Able to give signed informed consent
5. BMI 27-45 kg/m2, inclusive 6. Eligible male and female subjects must agree not to participate in a conception process (i.e. active attempt to become pregnant or to impregnate, egg or sperm donation, in vitro fertilization).
6. Considered to be in stable health in the opinion of the Investigator

Exclusion Criteria:

1. Prior participation in any study of lorcaserin.
2. Clinically significant new illness in the 1 month before screening
3. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol
4. History of any of the following cardiovascular conditions:

   * Myocardial infarction (diagnosed by cardiac enzyme[s] and/or diagnostic ECG), cerebral vascular accident (CVA), transient ischemic attack (TIA) or reversible ischemic neurologic deficit (RIND) within 6 months of screening
   * Cardiac arrhythmia requiring initiation of new medical or surgical treatment within 6 months of screening (stable medical therapy for > 6 months, pacemakers and/or defibrillators implanted > 6 months prior to screening are acceptable)
   * Unstable angina
   * History of pulmonary artery hypertension
5. Positive result of HIV, hepatitis B or hepatitis C screens
6. Initiation of a new prescription medication within 1 month prior to screening with the following exceptions:
7. Use of SSRIs, SNRIs, and other medications must meet washout period.
8. Participated in any clinical study with an investigational drug, biologic, or device within 1 month prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare the single-dose pharmacokinetic (PK) parameters of lorcaserin in the obese or overweight Elderly (> 65) to those obtained from the obese or overweight Adult (18-65)

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single oral dose of lorcaserin in obese or overweight Elderly (> 65) subjects and obese or overweight Adult (18-65) subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- CRI Worldwide - Lourdes Hospital, Willingboro, New Jersey, United States

REFERENCES:
- [Derived] Christopher RJ, Morgan ME, Tang Y, Anderson C, Sanchez M, Shanahan W. Pharmacokinetics and Tolerability of Lorcaserin in Special Populations: Elderly Patients and Patients with Renal or Hepatic Impairment. Clin Ther. 2017 Apr;39(4):837-848.e7. doi: 10.1016/j.clinthera.2017.03.004. Epub 2017 Mar 30. PMID 28365033